CLINICAL TRIAL: NCT06518629
Title: Photobiomodulation Before or After In-office Tooth Whitening for Sensitivity Reduction: a Blinded, Randomized, Controlled Study
Brief Title: Photobiomodulation Before or After Tooth Whitening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Dra, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universidade Federal do Pará
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Tooth Sensitivity; Tooth Bleaching; Laser Therapy
MeSH Terms: conditions — Dentin Sensitivity | interventions — Low-Level Light Therapy; Tooth Bleaching

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Only in-office tooth whitening will be performed. Patients will not undergo additional treatments, however, a simulation of the application of FBM will be performed before and after each CD session. The low-power laser (Therapy EC, DMC, São Carlos, SP, Brazil) will be positioned perpendicularly, in contact, over the cervical and apical region of each tooth included in the whitening treatment. During the simulation, the equipment will not be activated, that is, irradiation will not be carried out.
  Interventions: Other: Photobiomodulation with low power laser
- FBM-Before (Experimental): Low power laser will be used immediately before CD. The energy supplied to each tooth will be 4J, using infrared light (IF) at 808 nm (± 10 nm) at two perpendicular points (located in the apical and cervical region) on the buccal surface of the incisors, canines and premolars. The laser will be operated in continuous mode and an energy of 2J will be applied to each point. The protocol that will be used to treat tooth sensitivity was recommended by the equipment manufacturer. Immediately after each whitening treatment session, a FBM simulation will be performed, in the same way as described for the Placebo group.
  Interventions: Other: Photobiomodulation with low power laser
- FBM-After (Experimental): The low-power laser will be used immediately after tooth whitening. The FBM protocol will occur in the same way as described for the FBM-Before group. The FBM simulation will occur before the CD session begins and will occur in the same way as described for the Placebo group.
  Interventions: Other: Photobiomodulation with low power laser

INTERVENTIONS:
Other: Photobiomodulation with low power laser — All groups will undergo in-office whitening treatment with 35% hydrogen peroxide (Whitness HP, FGM, Joinville, SC, Brazil). Three whitening sessions will be carried out, considering a seven-day interval between sessions.
  Other Names: Tooth Bleaching

SUMMARY:
The objective is to evaluate the effect of photobiomodulation (PBM) applied before or after in-office tooth whitening in reducing tooth sensitivity (TS) and color change. Sixty-six patients aged between 18 and 28 years old, of both sexes, with good oral and general health will be selected for the study. A randomization process will be carried out to allocate participants into the three different groups: FBM-Before, FBM-After and Placebo. All groups will undergo in-office whitening treatment with 35% hydrogen peroxide (Whitness HP, FGM, Joinville, SC, Brazil). Three whitening sessions will be carried out, considering a seven-day interval between sessions. TS will be measured using a visual analogue scale (VAS) and a five-point numerical rating scale (NRS), while shade change will be assessed using a spectrophotometer: before the bleaching treatment (T0), after the first (T1), second (T2). ) and third (T3) weeks of treatment and 30 days (T4) after the end of the bleaching treatment.

DETAILED DESCRIPTION:
Ethical Considerations This research project will adhere to the recommendations of CONSORT (Consolidated Standards of Reporting Trials) (Turner et al., 2012). Participants will be fully informed about the risks, methods, and objectives of this study, and their participation will require the signing of a free and informed consent form (ICF), in accordance with the Declaration of Helsinki (World Medical Association, 2013).

All collected data will be used exclusively for scientific purposes, and the identity of the participants will remain confidential. Participation in the study may be withdrawn at any time, and confidentiality will be assured even in the event of treatment discontinuation.

Sample Size Calculation The sample size for this study was determined using GPower 3.1 (Heinrich-Heine-Universität Düsseldorf, Germany). The calculation was based on a prior study by Moosavi et al. (2016), which employed a methodology similar to that proposed in this investigation. The sample size was calculated with a statistical power of 80%, an alpha error of 5%, and a predicted dropout rate of 20%. The resulting sample size for this study is 22 patients per group.

Study Design The clinical study will be a randomized, parallel, double-blind, placebo-controlled trial. Randomization will be performed to allocate participants into three different groups: PBM-Before, PBM-After, and Placebo.

All groups will undergo in-office whitening treatment with 35% hydrogen peroxide (Whiteness HP, FGM, Joinville, SC, Brazil). Three whitening sessions will be performed, with a seven-day interval between sessions.

Sample Selection A total of 66 patients aged 18 to 28 years, of both genders, with good general and oral health, will be selected for the study. The right maxillary canine must be classified as shade A2 or darker, according to the Vita Classical shade guide (VITA Zahnfabrik, Bad Säckingen, Germany).

Individuals presenting with active caries or periodontal disease, visible cracks in anterior teeth, obvious malocclusion, restorations or prosthetics in anterior teeth, gastroesophageal disorders, severe internal tooth discoloration (due to tetracycline, fluorosis, or non-vital teeth), dentin exposure in anterior or posterior teeth, parafunctional habits, dental sensitivity, previous whitening treatment, or orthodontic treatment will be excluded. Additionally, pregnant or breastfeeding individuals will not be included in this study.

All participants will undergo prophylaxis using a rubber cup and pumice seven days prior to the start of the study and will receive oral hygiene kits to standardize the use of toothpaste without desensitizing agents.

Randomization and Allocation Concealment A collaborator, who will not participate in the clinical intervention stages of the study, will be responsible for the randomization process. Each participant's clinical record will be stored in coded envelopes to maintain allocation concealment during randomization. This process will be carried out using Random Allocation Software 1.0.0 (University of Medical Sciences, Isfahan, Iran), where an interval system will be generated for subject allocation into one of the three study groups.

Blinding To ensure blinding of study participants, efforts will be made to prevent them from seeing the light or hearing the sound of the laser device. The sound emitted by the laser during light emission will be simulated using the iTalk Recorder app (Griffin Technology, Nashville, Tennessee, USA) for iPhone 12 (Apple, Cupertino, CA, USA) (Pompeu et al., 2021). In addition, participants will wear headphones with a playlist to block any sound emitted by the laser device. All participants will wear protective glasses provided by the manufacturer during the PBM sessions. The operators will not be blinded, as they will need to activate the laser when necessary. However, the evaluators will remain unaware of group allocation.

Clinical Protocol

1. Photobiomodulation

   Participants will receive treatment based on their allocated group:

   Placebo (n=22): Only in-office whitening will be performed. Patients will not undergo additional treatments; however, a simulation of PBM application will be conducted before and after each whitening session. The low-power laser (Therapy EC, DMC, São Carlos, SP, Brazil) will be positioned perpendicularly, in contact with the cervical and apical regions of each tooth included in the whitening treatment. During the simulation, the device will not be activated, meaning no irradiation will be applied.

   PBM-Before (n=22): Low-power laser therapy will be used immediately before the whitening session. Energy of 4J will be delivered to each tooth using an infrared light (IF) at 808 nm (± 10 nm) at two perpendicular points (located in the apical and cervical regions) on the buccal surface of the incisors, canines, and premolars. The laser will operate in continuous mode, and an energy of 2J will be applied at each point. The protocol for treating dental sensitivity will follow the manufacturer's recommendations. Immediately after each whitening session, a PBM simulation will be performed as described for the Placebo group.

   PBM-After (n=22): The low-power laser will be applied immediately after the whitening treatment. The PBM protocol will be the same as described for the PBM-Before group. The PBM simulation will occur before the whitening session begins, as described for the Placebo group.
2. Dental Whitening For the whitening treatment, a gingival barrier will be placed using a light-curing resin (Top Dam, FGM, Joinville, SC, Brazil), followed by the application of a 35% hydrogen peroxide gel (Whiteness HP, FGM, Joinville, SC, Brazil). As per the manufacturer's instructions, three applications of the whitening gel will be made on the buccal surface of the incisors, canines, and premolars of both the upper and lower arches, each lasting 15 minutes, for a total of 45 minutes in each whitening session. The whitening treatment will consist of three sessions with a seven-day interval between them.

Post-Operative Sensitivity Assessment Participants will be instructed to complete a form (Appendix I) to record dental sensitivity based on individual pain perception. This form will be provided after each whitening session and returned at the next appointment, i.e., one week after each whitening session. Participants will record the intensity of pain at the following time intervals: (1) during the treatment; (2) up to 1 hour after each whitening session; (3) between 1 and 24 hours after each session; (4) between 24 and 48 hours; and (5) between 48 and 72 hours.

Participants will receive detailed instructions on how to complete the form. The evaluation form will include two pain scales: a five-point numeric rating scale (NRS) and a visual analog scale (VAS). For the NRS, participants will be asked to indicate a numerical value representing the degree of sensitivity, where 0 means no sensitivity, 1 mild, 2 moderate, 3 considerable, and 4 severe sensitivity.

For the VAS, a 10 cm horizontal line with scores of 0 and 10 at each end will be used, where 0 indicates no sensitivity and 10 indicates severe dental sensitivity. Participants will be instructed to mark the intensity of dental sensitivity with a vertical line along the horizontal scale each day. The distance in millimeters from the zero point will later be measured using a millimeter ruler to determine the level of pain intensity.

Color Evaluation The same researcher responsible for the clinical intervention will perform the color evaluation at four time points: baseline (T0), one week after the first whitening session (T1), one week after the second whitening session (T2), and 30 days after the end of treatment (T3). Color measurement will be performed using the VITA Easyshade spectrophotometer (VITA Zahnfabrik, Bad Säckingen, Germany), with the area of interest being the middle third of the buccal surface of the right maxillary canine.

To standardize the color readings, silicone guides (Cub Kit Profle, Vigodent) will be fabricated. For each canine, a window will be created on the buccal surface of the silicone guide using a metallic device with a 6 mm radius, matching the diameter of the spectrophotometer tip. The device's tip will be inserted into the silicone guide to obtain the color parameters of the CIELab* system, where L* represents lightness (light or dark); a* measures red (positive) or green (negative); and b* measures yellow (positive) or blue (negative) (Commission Internationale De L'Eclairage, 1978). The sum of the values measured for the upper canines will be used to calculate the average for each Lab* coordinate for each patient. ΔL*, Δa*, and Δb* will be calculated as the difference between the time intervals. The color difference between the baseline and the respective post-whitening time points will be calculated using the CIELab* (ΔE*ab)74 and CIEDE2000 (ΔE00) formulas (Luo et al., 2001; Della Bona et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes, in good oral and general health.
* The upper right canine should be classified as color A2 or darker, according to the Vita Classical scale (VITA Zahnfabrik, Bad Sackingen, Germany).

Exclusion Criteria:

* Active caries or periodontal disease
* Visible cracks in upper or lower anterior teeth
* Evident malocclusion, restorations and prosthetics in anterior teeth
* Gastroesophageal disorders
* Severe internal discoloration of the tooth (tetracycline, fluorosis or pulped teeth)
* Exposure dentin in anterior and/or posterior teeth
* Parafunctional habits
* Tooth sensitivity, previous bleaching treatment or orthodontic treatment
* Pregnant or breastfeeding women

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Tooth sensitivity | 21 days
  To assess pain sensitivity, patients will be instructed to fill out a form to record tooth sensitivity, based on individual pain perception. This form will be delivered at each whitening session, and will be returned to the researcher at the next appointment, that is, always one week after each whitening session.

SECONDARY OUTCOMES:
Color change | 51 days
  To measure shade, the VITA Easyshade spectrophotometer (VITA Zahnfabrik, Bad Säckingen, Germany) will be used, where the area of tooth correspondence to be evaluated will be the middle third of the buccal surface of the upper right canine. To standardize color readings, silicone guides will be made (Cub Kit Profle, Vigodent).

CONTACTS AND LOCATIONS:
Locations (1):
- Elma Vieira Takeuchi, Belém, Pará, Brazil